CLINICAL TRIAL: NCT05349526
Title: Anatomical Relationship Between Carotid Artery and Hyoid Bone in Stenotic and Non-stenotic Carotids: a Cohort Study of Symptomatic and Asymptomatic Carotid Endarterectomy Patients
Brief Title: Anatomical Relationship Between Carotid Artery and Hyoid Bone in Stenotic and Non-stenotic Carotids
Acronym: CAROTHYD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2022/DR-01
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2023-05

CONDITIONS: Stenoses, Carotid; Stroke
Keywords: computed tomography; carotid; atherosclerotic; plaque; density; stroke
MeSH Terms: conditions — Carotid Stenosis; Stroke; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stenotic carotid: patients with a stenotic carotid
  Interventions: Other: None, pure observational study
- non stenotic carotid: patients with non stenotic carotid
  Interventions: Other: None, pure observational study

INTERVENTIONS:
Other: None, pure observational study — None, pure observational study

SUMMARY:
Ischaemic stroke is attributable to thromboembolism caused by carotid atherosclerotic disease in 18-25% of patients. Guidelines for prevention of stroke (especially carotid endarterectomy) in patients with carotid atherosclerotic plaque are based on the quantification of the degree of stenosis.

The hyoid bone, in proximity to the carotid artery, has been implicated in the pathophysiology of carotid artery dissection, atherosclerotic carotid disease, and compressive syndromes. In atherosclerotic carotid disease, pressure on the carotid artery induced by these bone structures has been proposed to play a possible role in plaque formation and rupture, leading to stenosis, occlusion, or artery-to-artery embolism. In a recent ultrasound study, dynamic displacement of the carotid artery with interference of the hyoid bone during swallowing, named as "flip-flop" phenomenon (FFP) has been associated with carotid artery stenosis and stenosis-related stroke. Another study based on CTA assessment observed no association between hyoid-carotid distance and plaque thickness, stenosis, or progression of thickness/stenosis. In that study, in almost two-third of the patients CTA was performed for stroke/transient ischemic attack work-up, including a vast majority of patients with absence of carotid stenosis (median degree of carotid stenosis was 7%), and plaque-related stroke was not assessed.

The objective of this study is to determine the anatomic hyoid-carotid interaction (ie, hyoid-carotid distance, carotid position relative to the hyoid bone, and hyoid morphology) based on CTA and its relation to the degree of carotid stenosis and stenosis-related stroke.

ELIGIBILITY:
* Patients followed at the University Hospital of Nîmes between November 2016 and March 2020
* Age > 18 years
* Patients who underwent carotid endarterectomy for symptomatic or asymptomatic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of preoperative CTA of 206 consecutive adult patients (>18 years of age) who underwent carotid endarterectomy for symptomatic or asymptomatic stenosis, registered in the stroke database between November 2016 and March 2020 in Nîmes University Hospital (France).
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Distance hyoid-carotid artery | Base line, Day 0
  the closest distance between the hyoid bone and the outer vessel wall of the carotid artery(mm)
Carotid artery portion closest to the hyoid bone | Base line, Day 0
  Depending on the level of the carotid bifurcation: common carotid artery [CCA], carotid bifurcation [CB], or internal carotid artery [ICA])
Carotid artery position in regard to ipsilateral greater horn of the hyoid | Base line, Day 0
  The position of the carotid artery in regard to the ipsilateral greater horn of the hyoid (expressed in angle degree, with 0 to 90° corresponding to the posterolateral carotid position, 90 to 180° to anterolateral, 0 to -90° to posteromedial position, and -90 to-180° to anteromedial carotid position)
Hyoid bone morphology | base line, day 0
  Hyoid width (HW), hyoid length (HL), and hyoid circumferential length (HCL)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Salaun-Penquer E, Laurent-Chabalier S, Trandafir C, Cosma C, Parvu T, Wacongne A, Thouvenot E, Renard D. Relationship between hyoid-carotid distance, hyoid position and morphology and degree of stenosis and associated stroke: Hyoid-carotid relationship. J Stroke Cerebrovasc Dis. 2025 Jan;34(1):108106. doi: 10.1016/j.jstrokecerebrovasdis.2024.108106. Epub 2024 Nov 19. PMID 39571666